CLINICAL TRIAL: NCT05563142
Title: Venous Vascular Closure System Versus Manual Compression Following Single Shot Device AF Ablation - the Style-AF Study
Brief Title: Venous Vascular Closure System Versus Manual Compression Following Single Shot Device AF Ablation
Acronym: Style-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Prof. Roland Richard Tilz, Clinical Professor, Head of Rhythmology, University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Style-AF
Record Dates: First submitted 2022-09-27; First posted 2022-10-03 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Perclose ProStyle closure (Experimental): 50 patients treated with Perclose ProStyle suture-mediated closure device to achieve hemostasis
  Interventions: Procedure: deploying vascular closure device versus manual compression
- Group manual compression (Active Comparator): 50 patients treated with manual compression and one figure of eight suture
  Interventions: Procedure: deploying vascular closure device versus manual compression

INTERVENTIONS:
Procedure: deploying vascular closure device versus manual compression — patients will be randomized to either group 1 or group 2 in a 1:1 ratio:

SUMMARY:
Prospective, randomized, controlled, multi-center study to compare the safety and efficacy of the Perclose ProStyle suture-mediated closure device (PPS) as to manual compression (MC) for venous hemostasis following single shot device (SSD) based pulmonary vein isolation (PVI).

DETAILED DESCRIPTION:
The aim of this study is to show that the time to ambulation after PVI can be reduced by deploying vascular closure device versus manual compression and a figure-of-8 suture only. Safety, efficacy and feasibility of the PPS device should be proven, too.

ELIGIBILITY:
Inclusion Criteria:

* Patients age >18
* Elective catheter ablation for atrial fibrillation using a 6 to 14 Fr inner diameter introducer sheath with a minimum of 1 and maximum of 2 femoral venous access sites

Exclusion Criteria:

* Active systemic or cutaneous infection, or inflammation in vicinity of the groin
* Platelet count < 100,000 cells/mm3
* BMI > 45 kg/m2 or < 20 kg/m2
* Attempted femoral arterial access or inadvertent arterial puncture
* Procedural complications that interfered with routine recovery, ambulation, or discharge times
* Incorrect sheath placement
* Intraprocedural bleeding or thrombotic complications
* Access site-specific eligibility criteria to exclude problems with gaining access or location of sheath

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Time to ambulation | 6 hours
  elapsed time between removal of the final closure device or removal of the final sheath and when the patient can stand and walk 20 ft without evidence of venous re-bleeding from the femoral access site.

SECONDARY OUTCOMES:
total post procedure time | 6 hours
  elapsed time between removal of the last procedural device for the index procedure and when the patient was able to successfully ambulate
time to hemostasis | 6 hours
  elapsed time between removal of the closure device or the sheath and first observed and confirmed venous hemostasis, for each access site
time to discharge eligibility | 3 days
  elapsed time between removal of the final closure device or final sheath and when the patient was eligible for hospital discharge based solely on the assessment of the access site, as determined by the medical team
time to discharge | 3 days
  elapsed time between removal of the final closure device or final sheath and when the patient was discharged from the institution
time to closure eligibility | 6 hours
  elapsed time between removal of the last procedural device for the index procedure and removal of the first closure device or first sheath
Incidence of major adverse events | 30 days
  Incidence of major adverse events within 30 days after the procedure
Incidence of minor adverse events | 30 days
  Incidence of minor adverse events within 30 days after the procedure
Time to final hemostasis | 3 days
  Attainment of final hemostasis at all venous access sites and freedom from major venous access site closure-related complications

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen, North Rhine-Westphalia
  - Klinik für Innere Medizin III, Kiel, Schleswig-Holstein
  - Klinik für Rhythmologie, Lübeck, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: Undecided